CLINICAL TRIAL: NCT01115686
Title: Which Place for Branched-chain Aminoacids in the Treatment of Sleep Apnea Syndromes?
Brief Title: Branched-chain Aminoacids in Sleep Apnea Syndromes (ARSAS)
Acronym: ARSAS
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: I08024
Record Dates: First submitted 2010-04-30; First posted 2010-05-04 (Estimated); Last update posted 2018-08-22 (Actual); Status verified 2010-04

CONDITIONS: Sleep Apnea
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Branched-chain aminoacids (Active Comparator): Branched-chain aminoacids are natural constituents of the food. Branched-chain aminoacids will be orally administered in the form of capsules.
  Interventions: Drug: Branched-chain aminoacids
- placebo (Placebo Comparator): The placebo will be orally administered in the form of capsules
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Branched-chain aminoacids — Branched-chain aminoacids will be orally administered in the form of capsules, at the rate of a capsule for physical 7 Kilograms weighty and a day. Every capsule containing 375 milligrams of branched-chain aminoacids.
  The treatment will last 3 weeks.
  Arms: Branched-chain aminoacids
Drug: Placebo — Placebo will be orally administered in the form of capsules, at the rate of a capsule for physical 7 Kilograms weighty and a day.
  The treatment will last 3 weeks.
  Arms: placebo

SUMMARY:
The initial hypothesis is that branched-chain aminoacids (BCAA) administration could be beneficial to patients suffering from sleep apnea syndrome (SAS), the aim of the present work is to verify this hypothesis.

The literature data demonstrate that a BCAA complementation improves the physical performances, protects lean mass and increases VO2 max during training.

We demonstrated earlier that this complementation can cure at less partly the hypoxemia of chronic obstructive pulmonary patients by a stimulation of respiratory centres.

ELIGIBILITY:
Inclusion Criteria:

* Adult with healthy mind, who has attained his majority, and affiliated to Social Security.
* Patient suffering from SAS confirmed by polysomnography (PSG).
* Written informed consent form signed.

Exclusion Criteria:

* Patients receiving neuroleptics or benzodiazepines and affiliated drugs will not be included in the study.
* Patients suffering for severe SAS : those who have a number of IAH higher than 30 in a validated sleep hour, will be excluded for security reasons.
* Pregnant women, nursing mothers or women susceptible to procreate without efficient contraception.
* Patient presenting hypersensitivity to understudying products and their excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-06; Primary Completion 2012-06 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
The principal criterion of BCAA efficacy is based on the depth of arterial desaturation during sleep, assessed by the level of SaO2 during the validated sleep time measured during the polysomnography performed at the end of the study. | 2 years

SECONDARY OUTCOMES:
The secondary criteria are apnea and snore counting, the intergroup difference between the beginning and the end of treatment on nocturnal desaturations. | 2 years